CLINICAL TRIAL: NCT06419556
Title: Analgesic Efficacy of an Intermediate Cervical Plexus Block in Patients Undergoing Neck Surgeries. A Comparison Between Two Bupivacaine Concentrations.
Brief Title: Analgesic Efficacy of an Intermediate CPB in Neck Surgeries.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nagy Malak , MD, Lecturer of anesthesia ,SICU and pain, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-425-2023
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Thyroid; Neck; Bupivacaine
Keywords: Neck surgeries; Cervical Plexus Block; Bupivacaine
MeSH Terms: conditions — Thyroid Diseases | interventions — Cervical Plexus Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group H (Experimental): The patient's head was rested on a pillow and turned to the opposite side. A linear probe with higher frequencies was placed transversely over the midpoint of the SCM muscle. The carotid artery was identified and traced upwards to its bifurcation. Probe was then moved laterally to identify the tapering posterolateral end of the SCM muscle. Via an in-plane technique, a 22-gauge, 50 mm needle was advanced underneath the investing fascia of SCM muscle and above the interscalene groove until the "pop" on piercing the investing fascia was felt. Group H received 20 ml 0.25 % bupivacaine
  Interventions: Procedure: Cervical Plexus Block
- Group L received 20 ml 0.125% bupivacaine (Active Comparator): The patient's head was rested on a pillow and turned to the opposite side. A linear probe with higher frequencies was placed transversely over the midpoint of the SCM muscle. The carotid artery was identified and traced upwards to its bifurcation. Probe was then moved laterally to identify the tapering posterolateral end of the SCM muscle. Via an in-plane technique, a 22-gauge, 50 mm needle was advanced underneath the investing fascia of SCM muscle and above the interscalene groove until the "pop" on piercing the investing fascia was felt. Group L received 20 ml 0.125% bupivacaine.
  Interventions: Procedure: Cervical Plexus Block

INTERVENTIONS:
Procedure: Cervical Plexus Block — The patient's head was rested on a pillow and turned to the opposite side. A linear probe with higher frequencies was placed transversely over the midpoint of the SCM muscle. The carotid artery was identified and traced upwards to its bifurcation. the probe was then moved laterally to identify the tapering posterolateral end of the SCM muscle. Via an in-plane technique, a 22-gauge, 50 mm needle was advanced underneath the investing fascia of SCM muscle and above the interscalene groove until the "pop" on piercing the investing fascia was felt.

SUMMARY:
This study aims to investigate the analgesic efficacy of Intermediate Cervical Plexus Block combined with GA using two bupivacaine concentrations in patients undergoing neck surgeries (total thyroidectomy or total laryngectomy)

DETAILED DESCRIPTION:
This randomized comparative study was conducted in Cairo University hospitals after the approval of the institutional research and ethics committee. Informed consent was obtained from all participants. The Consolidated Standards of Reporting Trials (CONSORT) Guidelines were followed.

The patients were randomly allocated into two groups (H & L) using computer generated random numbers that were concealed in opaque envelopes. Group H received 20 ml 0.25 % bupivacaine and Group L received 20 ml 0.125% bupivacaine bilaterally.

* On arrival to the operating room, an 18G cannula was inserted with the infusion of 500 ml Ringer solution. Controloc 40 mg, ondansetron 8 mg, and dexamethasone 8 mg were administered as premedication. The diaphragmatic motion was assessed by a 3.5 MHz curvilinear transducer, siemens ACUSON X300 ultrasound. Each hemidiaphragm was first visualized by B-mode then M-mode was used to evaluate diaphragmatic excursion. For the right hemidiaphragm, the transducer was placed perpendicularly over the right subcostal margin in the anterior axillary line, the prob was then directed cephalad and dorsally to reach the posterior one-third of the diaphragm. Diaphragmatic excursions were measured and recorded in millimeters using the liver as an acoustic window during quiet breathing. The left hemidiaphragm was assessed in the same way using the spleen as an acoustic window.
* All patients connected to an electrocardiograph (ECG), pulse oximeter, and non-invasive blood pressure (NIBP), and baseline values of HR and MAP were measured and recorded. Additional monitoring in the form of a capnogram, invasive blood pressure (IBP) through a radial artery cannula, peripheral nerve stimulator (PNS), Bispectral index (BIS), and urine output were connected after induction of GA. Anesthesia was induced by intravenous fentanyl 2µg/kg, propofol 1.5-2 mg/kg, and atracurium 0.5 mg. When the TOF count showed the disappearance of T1 (0/4), an appropriate-size endotracheal tube was inserted and secured. Under complete aseptic conditions, ultrasound guided bilateral ICPB was performed by a single staff anesthetist who is skilled in carrying out regional anesthesia.
* ICPB technique: The patient's head was rested on a pillow and turned to the opposite side. A linear probe with higher frequencies was placed transversely over the midpoint of the SCM muscle. The carotid artery was identified and traced upwards to its bifurcation. the probe was then moved laterally to identify the tapering posterolateral end of the SCM muscle. Via an in-plane technique, a 22-gauge, 50 mm needle was advanced underneath the investing fascia of SCM muscle and above the interscalene groove until the "pop" on piercing the investing fascia was felt. The patient was then randomly allocated into two groups (H & L) using computer generated random numbers that were concealed in opaque envelopes. Group H received 20 ml 0.25 % bupivacaine and Group L received 20 ml 0.125% bupivacaine. The technique was repeated on the opposite side.
* During the intraoperative period, anesthesia was maintained with isoflurane 1.2-1.5 vol% to keep BIS value at 40-60 and atracurium 0.1mg/kg guided by PNS. Additional doses of fentanyl 0.05 µg/kg were administered when HR or MAP increased > 20% of the baseline values. MAP and HR were measured after the skin incision, and then every 30 minutes till the end of surgery. The failed block was considered when ≥ four additional doses of fentanyl were required to manage the increased MAP or HR after skin incision. At the end of the surgery, one gram of paracetamol plus 30 mg of ketorolac were administered.
* During the postoperative period, regular analgesia in the form of intravenous paracetamol one gram/8hr was prescribed. Pain severity was assessed by using the visual analog scale (VAS) (0= no pain and 100mm= worst pain) at 2, 4, 6, 8, 12, 18, and 24 hr postoperatively. Rescue analgesia in the form of intravenous morphine 0.05 mg/kg was given on the patient's complaint or when VAS ≥ 40 mm and repeated every 15-20 minutes until VAS < 40 mm with a maximum morphine dose of 40 mg per 24 hours. The duration of analgesia was calculated as the time elapsed from the end of the ICPB block procedure till VAS ≥ 40mm. The total postoperative morphine consumption over 24 hours was calculated. The measurement of diaphragmatic excursions was repeated as mentioned above, hemi-diaphragmatic paresis was divided into three grades, depending on the percentage of diaphragm movement compared with baseline to be: none (> 75%), partial paresis (25-75%), and complete paresis (< 25%)

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged ≥ 40 years
* ASA physical status I-III scheduled for total thyroidectomy or total laryngectomy under GA.

Exclusion Criteria:

* Patients with heart failure
* history of arrhythmias
* treatment with antiarrhythmic drugs
* impaired pulmonary
* Liver or kidney functions
* Neck infection or rash

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | duration of operation up to 6 hours
  duration of anesthesia and Block-skin incision time differ between two groups (two concentrations of bupivacaine)

SECONDARY OUTCOMES:
The diaphragmatic motions measured by M-mode ultrasonography | duration of operation up to 6 hours
  Measured at two-time points: before anesthesia (baseline) and on arrival to PACU, with the calculation of the hemi-diaphragmatic paresis depending on the percentage of diaphragm movement compared with baseline as follows: none (> 75%), partial paresis (25-75%), and complete paresis (< 25%).
Total postoperative Morphine consumption. | 24 hours
  Total postoperative Morphine consumption.
The postoperative VAS score | 24 hours
  scale (0= no pain and 100 mm= worst pain) and measured at 2, 4, 6, 8, 12, 18, and 24 hr postoperatively. Rescue analgesia in the form of intravenous morphine 0.05 mg/kg given on the patient's complaint or when VAS ≥ 40 mm and repeated every 15-20 minutes until VAS < 40 mm with a maximum morphine dose of 40 mg per 24 hours.
Hemodynamics | duration of operation up to 6 hours
  Intraoperative MAP and HR were measured after the skin incision, and then every 30 minutes until the end of surgery.
opioid consumption. | duration of operation up to 6 hours
  Intraoperative opioid (fentanyl) consumption.The failed block was considered when ≥ four additional doses of fentanyl were required to manage the increased MAP or HR after skin incision.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Hospitals. kasralainy, Cairo, Governorate, Egypt